CLINICAL TRIAL: NCT00542035
Title: A RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL-GROUP ANALGESIC EFFICACY TRIAL OF ORAL ARRY-371797 IN SUBJECTS UNDERGOING THIRD MOLAR EXTRACTION
Brief Title: A Study of ARRY-371797 in Subjects Undergoing Third Molar Extraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ARRAY-797-221; C4411008 (Other: Alias Study Number)
Record Dates: First submitted 2007-10-05; First posted 2007-10-10 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Dental Pain
Keywords: Analgesia
MeSH Terms: conditions — Toothache; Agnosia | interventions — ARRY-371797

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ARRY-371797 (Experimental)
  Interventions: Drug: ARRY-371797, p38 inhibitor; oral
- Placebo, ARRY-371797 (Experimental)
  Interventions: Drug: Placebo; oral; Drug: ARRY-371797, p38 inhibitor; oral
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; oral

INTERVENTIONS:
Drug: ARRY-371797, p38 inhibitor; oral — dose 1, dose 2
  Arms: ARRY-371797
Drug: Placebo; oral — dose 1, dose 2
  Arms: Placebo
Drug: Placebo; oral — dose 1
  Arms: Placebo, ARRY-371797
Drug: ARRY-371797, p38 inhibitor; oral — dose 2
  Arms: Placebo, ARRY-371797

SUMMARY:
This is a Phase 2 study designed to test the ability of investigational study drug ARRY-371797 to reduce pain either perioperatively or postoperatively in a third molar extraction pain model, and to further evaluate the drug's safety. Approximately 150 subjects from the US will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Scheduled for outpatient oral surgical procedure to remove 2 ipsilateral third molars, at least 1 of which is mandibular and fully or partially impacted by bone.
* Females of childbearing potential must be willing to use an acceptable method of contraception within 14 days prior to first dose of study drug until the completion of the follow-up procedures.
* Body weight >50 kg (110 lbs).
* Good health determined by medical history, physical examination, vital signs and clinical laboratory results of non-clinical significance.
* Additional criteria exist.

Key Exclusion Criteria:

* Positive urine drug screen.
* Use of prescription or nonprescription drugs, herbal or dietary supplements, vitamins, or grapefruit juice within 14 days prior to first dose of study drug.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2007-11-11 (Actual); Primary Completion 2008-02-11 (Actual); Study Completion 2008-02-11 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of the study drug dosed either perioperatively or postoperatively in terms of total pain relief (TOTPAR) and total pain intensity (visual analog scale, VAS). | 6 hours post dose 2
Characterize the safety profile of the study drug in terms of adverse events, clinical laboratory tests, electrocardiograms and vital signs. | Duration of study

SECONDARY OUTCOMES:
Compare the efficacy of the study drug dosed perioperatively versus postoperatively in terms of total pain intensity (VAS). | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - SCIREX Research Center, San Marcos, Texas
  - SCIREX Research Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests